CLINICAL TRIAL: NCT03755336
Title: Variability and Specificity in Reactive Stabilization Movements to Diverse Slip Perturbations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 0877-18-EP; 2P20GM109090-06 (NIH)
Record Dates: First submitted 2018-11-21; First posted 2018-11-27 (Actual); Results first posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Slip Perturbations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Slipping Perturbations (Experimental): Participants will be exposed to a series of 12 unannounced slip perturbations while walking overground. These perturbations will be delivered at 3 different times within the gait cycle - early phase, middle phase, and late phase.
  Interventions: Other: Administered Slip Perturbations

INTERVENTIONS:
Other: Administered Slip Perturbations — Participants will be exposed to a series of 12 unannounced slip perturbations while walking overground. These perturbations will be delivered at 3 different times within the gait cycle - early phase, middle phase, and late phase.

SUMMARY:
Recent research on slips has shown that use of perturbation training to improve specific motor skills to resist slips can vastly reduce falls. However, these interventions have only addressed slips occurring at heel-strike, and not the diverse range of slipping disturbances presented by a complex environment. This project will focus on slips that occur across the gait cycle, and the reactive stabilization movements that follow.

Participants from two age groups will be enrolled: younger (19 - 35 years of age) and older (65-79 years of age). Each participant will participate in 3 visits within the span of 1 week. On the initial visit, participants will perform informed consent, have demographic and body measurement information collected and complete medical and physical activity questionnaires. Upper and lower body strength will be measured using a hand-held dynamometer during the first and last visits. On each of the three visits, subjects will perform a gait variability assessment followed by a diverse slip perturbation assessment. Participants will complete four slips in each of early, middle, and late stance on each visit. Measures of falls, slip severity, and reactive stabilization movements will be calculated.

DETAILED DESCRIPTION:
Recent research on slips has shown that use of perturbation training to improve specific motor skills to resist slips can vastly reduce falls. However, these interventions have only addressed slips occurring at heel-strike, and not the diverse range of slipping disturbances presented by a complex environment. This study will focus on slips that occur across the gait cycle, and the reactive stabilization movements that follow. Slips at different phases of the gait cycle have unique biomechanical contexts, and successful reactive stabilization movements are likely to be highly specific to that context. Yet nothing is known about the specificity of the repertoire of reactive stabilization movements to resist different slip conditions. Furthermore, variability in the repertoire of reactive stabilization movements is likely to affect the success/failure rate of resisting these disturbances. Thus, the objective of the proposed study is to determine the roles of variability and specificity in reactive stabilization movements to resist falling in diverse slipping conditions.

A novel wearable apparatus for slipping perturbations (WASP) will deliver lifelike, unexpected slips in early, middle and late stance in younger (19 - 35 years of age) and older adults. Biomechanical analysis based on three-dimensional motion capture data of the reactive stabilization movements will generate novel results on the specificity and variability of protective stepping and arm swinging responses. The central hypothesis is that increases in specificity and decreases in variability of reactive stabilization movements will reduce fall rates. The long-term objective of this research is to support future studies into the repertoire of reactive stabilization movements across the full range of disturbances faced in navigating the environment.

Each participant will participate in 3 visits within the span of 1 week. On the initial visit, participants will perform informed consent, have demographic and body measurement information collected and complete medical and physical activity questionnaires. Upper and lower body strength will be measured using a hand-held dynamometer during the first and last visits. On each of the three visits, subjects will perform a gait variability assessment followed by a diverse slip perturbation assessment. Before recording data, retroreflective markers will be placed on specific anatomical locations. These locations are defined to create a full-body dynamics model. For gait variability assessment, participants will be familiarized with the activity, then they will walk on a treadmill for 5 minutes at a prescribed pace of 1.3 meters per second while whole body kinematics are collected. Both linear and nonlinear measures of gait variability will be calculated to determine possible relationships between these measures and other outcome variables such as learning rate for reactive movements and fall rate.

For diverse slip perturbation assessment, participants will walk overground back and forth across a large motion capture area. Previous studies show that walking speed is highly correlated with some outcome measures, specifically variations in whole body angular momentum, gait variability measures, and loss of balance following a slip. Therefore, gait speed will be controlled to 1.3 ± 0.2 m/s, a typically comfortable speed for both younger and older adults. Participants will be informed that a slip may occur, and that if slipped, they should attempt to maintain balance and continue walking. Participants will then be slipped without warning at a randomly chosen time after 1 to 3 minutes of walking. Slips will be administered to both feet simultaneously during early, middle or late stance in a randomized order. After each slip, participants will rest seated for 5 minutes. During this rest period, motion capture data and force data from the harness will be recorded, and the WASP will be reset for the next trial. Participants will complete four slips in each of early, middle, and late stance on each visit. Measures of falls, slip severity, and reactive stabilization movements will be calculated.

ELIGIBILITY:
Inclusion Criteria:

* Age 19-35 years for younger adults group, or age 65-79 years for older adults group.

Exclusion Criteria:

* Uncontrolled hypertension
* Peripheral arterial disease
* Vertigo
* Meniere's disease
* Chronic dizziness
* History of back or lower extremity injury
* Surgery that affects the subject's mobility
* Any neurological disease or impairment that affects limits the ability to walk, e.g. Stroke, Parkinson's disease, Multiple sclerosis

Ages: 19 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nathaniel H Hunt, PhD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska-Omaha, Biomechanics Research Building, Omaha, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Slipping Perturbations - Younger Adults: The intervention involves exposing younger adult participants to a series of 12 unannounced slip perturbations while walking overground. These perturbations will be delivered at 3 different times within the gait cycle - early phase, middle phase, and late phase.
  Administered Slip Perturbations: Slips will be administered in early, middle or late phases of stance during overground walking.
- Slipping Perturbations - Older Adults: The intervention involves exposing older adult participants to a series of 12 unannounced slip perturbations while walking overground. These perturbations will be delivered at 3 different times within the gait cycle - early phase, middle phase, and late phase.
  Administered Slip Perturbations: Slips will be administered in early, middle or late phases of stance during overground walking.
Period: Overall Study
Arm/Group | Slipping Perturbations - Younger Adults | Slipping Perturbations - Older Adults
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Slipping Perturbations - Younger Adults | Slipping Perturbations - Older Adults | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 0 | 22
  >=65 years | 0 | 22 | 22
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 11 | 21
  Male | 12 | 11 | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 21 | 22 | 43
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 6 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 15 | 22 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: centimeters] | 171.3 (15.2) | 169.9 (11.0) | 170.6 (13.0)
Weight [Mean (Standard Deviation); unit: kilograms] | 73.6 (12.8) | 81.3 (17.3) | 77.5 (15.6)

OUTCOME MEASURES:

1. Primary Outcome: Fall Rates
Description: Percentage of trials which result in a fall. Falls are classified when the maximum force on the load cell in the harness system exceeds 30% body weight.
Time Frame: Up to 7 days
Population: Participants were administered slips 12 times in a session for each of 3 sessions.
Measure: Number; unit: Percentage of trials resulting in falls.
Units Other Than Participants: Trials
Arm/Group | Slipping Perturbations - Younger Adults | Slipping Perturbations - Older Adults
Number analyzed (Participants) | 22 | 22
Number analyzed (Trials) | 792 | 792
Percentage of trials resulting in falls. | 18.3 | 16.0

2. Secondary Outcome: Total Heel Displacement of the Slipping Foot Following Slip Perturbation
Description: The total displacement of the slipping foot from the point of administered slip perturbation, until the foot stops sliding is assessed.
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

3. Secondary Outcome: Trunk Angular Momentum Following Slip Perturbation
Description: Angular momentum of the trunk is assessed during the period of time from the onset of slip perturbation until the subject recovers or falls.
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

4. Secondary Outcome: Position of the Recovery Step Following Slip Perturbation
Description: Position of the placement of the swing foot relative to the center of mass in the transverse plane following slip perturbation will be assessed.
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

5. Secondary Outcome: Coefficient of Variation of Stride Time Time Series
Description: The coefficient of variation of the time series of stride times during treadmill walking is assessed.
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

6. Secondary Outcome: Maximum Heel Sliding Velocity of the Slipping Foot Following Slip Perturbation
Description: The maximum velocity of the slipping foot will be assessed within the period from the administered slip perturbation, until the foot stops sliding.
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

7. Secondary Outcome: Time of the Recovery Step Following Slip Perturbation
Description: Time of the placement of the swing foot relative to the onset of the administered slip perturbation is assessed
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

8. Secondary Outcome: Sample Entropy of Stride Time Time Series
Description: The sample entropy of the time series of stride times during treadmill walking is assessed.
Time Frame: Up to 7 days
Reporting Status: Not Posted, anticipated posting 2026-12

ADVERSE EVENTS:
Time Frame: Up to 7 days
Description: This protocol was not expected to put participants at risk for Serious Adverse Events, or at risk for All-Cause Mortality.
Arm/Group | Slipping Perturbations - Younger Adults | Slipping Perturbations - Older Adults
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

LIMITATIONS AND CAVEATS:
Fall rates were derived from controlled walking trials using a safety harness on a sliding gantry. The harness may have influenced natural recovery responses. Additionally, laboratory conditions and participants' awareness of slip risk could have induced anticipatory behaviors, limiting generalizability.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03755336/Prot_SAP_000.pdf
  • Informed Consent Form (2023-02-09): https://cdn.clinicaltrials.gov/large-docs/36/NCT03755336/ICF_001.pdf